CLINICAL TRIAL: NCT07144007
Title: Van Yuzuncu Yil University Faculty of Medicine Ethics Committee
Brief Title: Prevention of Emergence Agitation in Rhinoplasty With Subanesthetic Propofol and Single-Dose Dexmedetomidine: A Prospective Double-Blind Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Mehmet Emin Keskin, assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025/04-07
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Emergence Agitation
Keywords: emergence agitaion; Propofol; Dexmedetomidine; Rhinoplasty
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Intervention Model Description: 80 patients scheduled for rhinoplasty will be randomly assigned to two groups. After nasal packing placement, one group will receive intraoperative 0.5 mg/kg propofol, while the other group will receive 10-minute infusion of 0.5 mcg/kg dexmedetomidine.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Group-D) (Active Comparator): Group-D: Dexmedetomidine group (n:40). In rhinoplasty, 10 minute infusion of 0,5 mcg/kg dexmedetomidine will be administered after nasal packing.
  Interventions: Drug: Dexmedetomidine
- Propofol (Group-P) (Experimental): Group-P: Propofol group (n:40). In rhinoplasty, 0,5 mg/kg propofol IV bolus will be administered after nasal packing.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — In rhinoplasty, 10 minute infusion of 0,5 mcg/kg dexmedetomidine will be administered after nasal packing
  Arms: Dexmedetomidine (Group-D)
Drug: Propofol — In rhinoplasty, 0,5 mg/kg propofol IV bolus will be administered after nasal packing
  Arms: Propofol (Group-P)

SUMMARY:
To compare of prevention of emergence agitation in rhinoplasty with subanesthetic propofol and single dose dexmedetomidine

DETAILED DESCRIPTION:
The study will have a double-blind design and will be conducted after obtaining an approval from the local ethics committee. The study will include 80 patients planned for elective rhinoplasty, aged 18-65 years with an ASA score of I-II. The patients will be randomized by sealed tender and will be divided into 2 groups with 40 patients each. All cases will receive routine preparation for general anesthesia. For anesthesia induction 0,03 mg/kg midazolam, 2 mcg/kg fentanyl, 2 mg/kg propofol and 0.6 mg/kg rocuronium will be used. Anesthesia will be maintained with 60% air, 40% oxygen and 1 MAC sevoflurane. If intraoperatively needed, an additional dose of 0.5 mcg/kg fentanyl and 0.15 mg/kg rocuronium will be administered. If necessary, nicardipine infusion will be administered to provide controlled hypotension. Before the end of the surgery, 15 mg/kg paracetamol and 1 mg/kg tramadol will be administered for postoperative analgesia. After the nasal tampons are placed, one group will receive 0.5 mg/kg propofol, and the other group will receive 0.5 mcg/kg dexmedetomidine IV infusion over 10 minutes. 4 mg/kg sugammadex will be administered as a muscle relaxant reversal agent. The patient will be extubated when spontaneous breathing occurs and the patient opens their eyes with verbal stimulation. Agitation status will be assessed with the Richmond Agitation Sedation Scale (RASS) at 1 minute after extubation. Heart rate, systolic, diastolic, mean arterial pressures and saturation values will also be recorded before and after anesthesia induction, at the 5th, 10th, 15th, 20th, 25th, 30th minutes after intubation, at the 1st, 5th, 10th and 15th minutes after extubation. Additionally, if meaningless head and hand-arm movements, laryngospasm, nausea-vomiting, hypoxia (SpO2: <85%) occur at the 1st, 5th, 10th and 15th minutes after extubation, they will be recorded. Also recovery time will be recorded. All data will be recorded and statistical analysis will be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for rhinoplasty
* Between 18-65 years
* ASA I-II group

Exclusion Criteria:

* Those who are outside the age range of 18-65
* Those who are ASA III and above
* Those with renal,hepatic, cardiac and respiratory diseases
* Those with a known allergy to the medication to be used
* Those who underwent urinary catheterization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Agitation status | 1. minute after extubation
  The effect on prevention of emergence agitation of propofol and dexmedetomidine will be evaluated by an anaesthetist with the Richmond Agitation Sedation Scale (RASS) at 1 minute after extubation

SECONDARY OUTCOMES:
Heart rate | perioperatively defined times
  Heart rate will be measured pre-induction of anesthesia, post-induction of anesthesia, 5th, 10th, 15th minutes after intubation, during extubation, 1st, 5th, 10th, 15th minutes after extubation
Blood Pressure | perioperatively defined times
  Systolic blood pressure, diastolic blood preesuure, mean arterial pressure will be measured pre-induction of anesthesia, post-induction of anesthesia, 1st, 5th, 10th, 15th minutes after intubation, during extubation, 5th, 10th, 15th minutes after extubation
oxygen saturation | perioperatively defined times
  Oxygen saturation will be measured pre-induction of anesthesia, post-induction of anesthesia, 5th, 10th, 15th minutes after intubation, during extubation, 1st, 5th, 10th, 15th minutes after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Şükran Sevimli, Assoc. Prof., Study Director — Yuzuncu Yil University
Locations (1):
- Van Yüzüncü Yıl University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol anda statistical analysis plan will be share with other researchers
Supporting Information: Study Protocol, SAP
Time Frame: 1 year
Access Criteria: The access can be provided via the e-mail addresses below emin6559@hotmail.com

REFERENCES:
- [Background] Makkar JK, Bhatia N, Bala I, Dwivedi D, Singh PM. A comparison of single dose dexmedetomidine with propofol for the prevention of emergence delirium after desflurane anaesthesia in children. Anaesthesia. 2016 Jan;71(1):50-7. doi: 10.1111/anae.13230. Epub 2015 Oct 7. PMID 26444149